CLINICAL TRIAL: NCT05280795
Title: an Audit on Postoperative Variations in Anemia Treatment After Major Gynecological Surgery
Brief Title: Audit on Anemia Variation After Major Gynacological Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yossra G. Rateb, principal investigator, Assiut University
Other Study IDs: anemia follow up
Record Dates: First submitted 2021-11-20; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to increase our understanding of variability in adherence to anaemia management guidelines and to assess the impact of anaemia management in clinical care following major gynaecological surgery

DETAILED DESCRIPTION:
Anemia affects nearly a quarter of the world and is common in surgical patients with a third of patients presenting with preoperative anemia and three quarters of patients discharged from hospital with anemia. The World Health Organization defines anemia as an insufficient circulating red cell mass, with haemoglobin (Hb) concentration of < 130 g.l-1 for men and < 120 g.l-1 for women .

Perioperative anemia is associated with increased postoperative complications and delayed patient recovery leading to increased post-operative morbidity and mortality. Anaemia also leads to an increased use of allogeneic blood transfusions, which is an independent risk for poorer patient outcomes.

Postoperative anemia can be due to blood loss at operation or secondary to the inflammatory process associated with surgery, which causes an increase in hepcidin production resulting in functional iron deficiency and reduced red cell production.

In recent years, there has been a significant increase in the use of intravenous iron therapy for preoperative anemia in line with major international guidelines

ELIGIBILITY:
Inclusion Criteria:

* Age: Adult, 18_60 years
* Procedure: A major gynecological surgery is defined as an operation with an incision into the abdominal cavity and anticipated duration of more than one hour. Procedures performed using any surgical approach, including open and laparoscopic surgery are included.
* Urgency: Patients undergoing planned (elective or expedited) or unplanned (emergency) surgery

Exclusion Criteria:

* Procedures: surgery classified as minor operations such as; diagnostic laparoscopy (emergency or elective), D&C.
* Indication: Palliative procedures as determined pre-operatively and explicitly stated in the medical record or consent form.
* Return to theatre: Each patient should only be included in the study once. Patients returning to theatre due to complications following earlier surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: any female 18 to 60 years undegoing major gynecological surgery
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
the rate of anemia after major gynecological surgery | one month
  percentage of patients with anemia after surgery

CONTACTS AND LOCATIONS:
Overall Officials: sayed mostafa, Study Director — Assiut University
Locations (1):
- Assuit university, Multiple Locations, Egypt

REFERENCES:
- [Background] Carson JL, Duff A, Poses RM, Berlin JA, Spence RK, Trout R, Noveck H, Strom BL. Effect of anaemia and cardiovascular disease on surgical mortality and morbidity. Lancet. 1996 Oct 19;348(9034):1055-60. doi: 10.1016/S0140-6736(96)04330-9. PMID 8874456
- [Background] McLean E, Cogswell M, Egli I, Wojdyla D, de Benoist B. Worldwide prevalence of anaemia, WHO Vitamin and Mineral Nutrition Information System, 1993-2005. Public Health Nutr. 2009 Apr;12(4):444-54. doi: 10.1017/S1368980008002401. Epub 2008 May 23. PMID 18498676